CLINICAL TRIAL: NCT06012513
Title: Sleep Disorders and Quality of Life in Patients With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Safwat Mahmoud Ahmed, Doctor, Assiut University
Other Study IDs: sleep disorders in MS
Record Dates: First submitted 2023-07-27; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To determine sleep disturbance in different types of multiple sclerosis.
2. To asses the effect of sleep disturbance on quality of life in patients with multiple sclerosis.
3. Correlation between sleep disturbance in different types of multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis(MS) is a neurodegenerative disease of the central nervous system that commonly affects young adults. The disease is characterized by neurological symptoms that may lead to long-term physical disability. Patients with MS have many other problems associated with their disease, as obstructive sleep apnea (OSA) that characterized by obstructions of the respiratory tract throughout the night leadind to wake up the patients many times to achieve the right muscle tone and receive adequate oxygenation. Most patients with MS complain from poor sleep.It may be due to pain, fatigue, depression and immunotherapy that have been considered as potential factors, which could have role in sleep disturbances among MS patients.Restless leg syndrome (RLS) may trigger sleep disorders, especially insomnia, in patients with MS. Patients with sleep disorders may complain excessive daytime sleepiness, impaired concentration, altered mood, and fatigue. they are at risk to develop other problems,as vascular diseases, obesity, and diabetes, which further threaten long-term health.So patients with MS have lower quality of life(QoL) than healthy ones. Multiple Sclerosis Quality of Life-54 (MSQoL-54) questionnaire is the most common and standardized disease-specific questionnaire that based on the generic SF-36 QoL instrument.

ELIGIBILITY:
Inclusion Criteria:

1. All patients fulfill the criteria of case definition of multiple sclerosis.
2. Gender: both sexes are included.
3. Willingness to participate in the study and to be subjected to the disease-related examinations and assessments.
4. Willing and able to provide informed consent.

Exclusion Criteria:

1. Patients unable to give informed consent.
2. Patients with history of psychiatric disorders or collagen disease such as Behcet's disease or other neurological or medical disease

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Multiple Sclerosis according to McDonald Criteria 2017 attending the neurology outpatient clinic, Department of Neurology and Psychiatry,Assiut University
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of different types of sleep disorders in patients with multiple sclerosis | Baseline
  Identification of different types of sleep disorders in patients with multiple sclerosis using different scales

REFERENCES:
- [Background] Tachibana N, Howard RS, Hirsch NP, Miller DH, Moseley IF, Fish D. Sleep problems in multiple sclerosis. Eur Neurol. 1994;34(6):320-3. doi: 10.1159/000117070. PMID 7851452
- [Background] Merlino G, Fratticci L, Lenchig C, Valente M, Cargnelutti D, Picello M, Serafini A, Dolso P, Gigli GL. Prevalence of 'poor sleep' among patients with multiple sclerosis: an independent predictor of mental and physical status. Sleep Med. 2009 Jan;10(1):26-34. doi: 10.1016/j.sleep.2007.11.004. Epub 2008 Jan 22. PMID 18207453